CLINICAL TRIAL: NCT04074590
Title: A Randomized, Multi-center, Subject and Investigator-blinded, Placebo-controlled, Parallel-group Study to Assess the Efficacy Safety and Tolerability of LYS006 in Patients With Mild to Moderate Ulcerative Colitis
Brief Title: Study of Efficacy, Safety, and Tolerability of LYS006, in Patients With Mild to Moderate Ulcerative Colitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision due to strategic considerations
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLYS006X2202; 2019-003113-34 (EudraCT Number)
Record Dates: First submitted 2019-08-29; First posted 2019-08-30 (Actual); Results first posted 2023-11-09 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Colitis, Ulcerative
Keywords: ulcerative colitis, efficacy, safety
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: This is a randomized, placebo-controlled, subject and investigator blinded, multicenter, non-confirmatory, parallel group, proof of concept study in patients with mild to moderate ulcerative colitis. This study consists of a screening period of up to 4 weeks, and a 8 week treatment period followed by a 30 day post treatment period safety follow up. The maximum study duration for each such including the 4 week screening period is 16 weeks.
  At the beginning of the treatment period, subjects will be randomized to one of the two following treatment groups in 2:1 ratio:
  * LYS006
  * matching placebo
Who Masked: Participant, Investigator
Masking Description: Subject and investigator blinded via randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LYS006 (Experimental): Experimental drug
  Interventions: Drug: LYS006
- Placebo (Placebo Comparator): Placebo comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LYS006 — capsule for oral use
  Arms: LYS006
Drug: Placebo — capsule for oral use
  Arms: Placebo

SUMMARY:
The purpose of the study was to assess preliminary efficacy, safety, and tolerability of LYS006 in adult patients with mild to moderate ulcerative colitis and to determine if LYS006 has an adequate clinical profile for further development in this indication.

DETAILED DESCRIPTION:
This was a randomized, placebo-controlled, subject and investigator blinded, multicenter, non-confirmatory, parallel group, proof of concept study in patients with mild to moderate ulcerative colitis. This study consisted of a screening period of up to 4 weeks, and a 8 week treatment period followed by a 30 day post treatment period safety follow up. The maximum study duration for each participant including the 4 week screening period was 16 weeks.

At the beginning of the treatment period, subjects were randomized to one of the two following treatment groups in 2:1 ratio

* LYS006
* matching placebo

ELIGIBILITY:
Key Inclusion Criteria:

* Male and female subjects 18-75 years of age with an established diagnosis of ulcerative colitis at least 3 months prior to screening are eligible for the study.
* Patients must have active disease with a full Mayo Score between 5 and 10 (inclusive) with an endoscopy score of 2 or 3; rectal bleeding and stool frequency scores 1 to 3 and a physician's global assessment of 1 or 2.
* Patients must have responded inadequately to conventional therapy with oral 5-ASA prior to screening.

Key Exclusion Criteria:

* Has previous diagnosis with Crohn's disease, indeterminate colitis, microscopic colitis or acute diverticulitis based on medical history.
* History of toxic megacolon, abdominal abscess, symptomatic colonic stricture, or stoma; history or is at risk of colectomy.
* Treatment with biologics within 3 months or 5 half-lives (whichever is longer) prior to screening endoscopy, non-biologics advanced therapies within 4 weeks prior to screening endoscopy, systemic immunosuppressant or immunomodulator within 6 week, topical treatment with 5-ASA or steroids within 2 weeks prior to screening endoscopy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-11-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- Novartis Investigative Site, Sofia, Bulgaria
- Czechia (2):
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Zlín, Czech Republic
- Novartis Investigative Site, Berlin, Germany
- Poland (3):
  - Novartis Investigative Site, Nowy Targ, Lesser Poland Voivodeship
  - Novartis Investigative Site, Warsaw, Masovian Voivodeship
  - Novartis Investigative Site, Poznan
- Novartis Investigative Site, Novosibirsk, Russia
- Novartis Investigative Site, Košice, Slovakia

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: Patient Lay Trial Summary — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1663

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 9 investigative sites in 6 countries.
Pre-assignment Details: After signing informed consent, screening evaluations took place from Day -28 to Day -1. During that period all safety and other assessments were performed to evaluate eligibility. Eligible patients returned for the Baseline visit on Day 1. Eligibility was confirmed prior to randomization and required baseline assessments were completed prior to dosing on Day 1.
Groups:
- LYS006 20mg: LYS006 20mg oral dose, twice daily
- Placebo: Placebo oral dose, twice daily
Period: Overall Study
Arm/Group | LYS006 20mg | Placebo
Started | 16 | 7
Completed | 12 | 7
Not Completed | 4 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LYS006 20mg | Placebo | Total
Number analyzed (Participants) | 16 | 7 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (12.20) | 45.7 (12.37) | 40.6 (12.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 8 | 2 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 16 | 7 | 23

OUTCOME MEASURES:

1. Primary Outcome: Clinical Remission Rate at the End of the Study Treatment
Description: The Mayo score is an instrument designed to measure activity of ulcerative colitis. The Mayo score comprises of four sub scores: stool frequency, rectal bleeding, endoscopic findings and the Physician's Global Assessment (PhGA). Each sub score is graded from 0 to 3 with higher scores indicating more severe disease. The full Mayo score is the sum of four sub scores, ranging from 0 to 12. Clinical remission is defined as a full Mayo score of 2 points or lower, with no individual subscore exceeding one point. The clinical remission rate is expressed as percentage of participants. The binary endpoint of clinical remission rate (Yes/No) at the EoT visit was modelled with binomial distribution and analyzed via the Bayesian approach with baseline total Mayo score and treatment group as explanatory variables, to compare the remission rates between the LYS006 and placebo groups.
Time Frame: Week 8
Population: The PD analysis set included all participants who received any study drug and had no protocol deviations with relevant impact on PD data.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | LYS006 20mg | Placebo
Number analyzed (Participants) | 14 | 7
Percentage of participants | 8.95 [0.87 to 23.31] | 12.24 [5.67 to 24.12]
Statistical Analysis 1: Comparison: LYS006 20mg vs Placebo; Test type: Other — A Bayesian analysis of clinical remission rate (based on total Mayo score) with binomial distribution, was modelled with baseline total Mayo score and treatment group as explanatory variables, to compare the remission rates between LYS006 and placebo groups; p = 0.314, Bayesian analysis — Posterior probability that clinical remission rate is better than placebo: Prob (diff>0); Posterior estimate treatment difference = -3.29, 90% CI 2-sided [-18.02 to 13.23] — 90% credible intervals are reported on the treatment difference
Statistical Analysis 2: Comparison: LYS006 20mg vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.037, Bayesian analysis — Posterior probability that clinical remission rate >15% over placebo: Prob (diff>0.15); Posterior estimate treatment difference = -3.29, 90% CI 2-sided [-18.02 to 13.23] — 90% credible intervals are reported on the treatment difference

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Number of participants with treatment emergent AEs, AEs led to study treatment discontinuation, SAEs and SAEs led to study treatment discontinuation.
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum duration of approximately 86 days.
Population: The safety analysis set included all participants that received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | LYS006 20mg | Placebo
Number analyzed (Participants) | 16 | 7
Participants
  At least one AE | 7 | 5
  At least one SAE | 0 | 0
  AE leading to discontinuation | 2 | 0
  SAE leading to discontinuation | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum duration of approximately 86 days
Groups:
- LYS006 20 mg: LYS006 20 mg oral dose, twice daily
- Total: Total
Arm/Group | LYS006 20 mg | Placebo | Total
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/7 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/7 | 0/23
Other Adverse Events (participants affected / at risk) | 7/16 | 5/7 | 12/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LYS006 20 mg (N=16) | Placebo (N=7) | Total (N=23)
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 1
Colitis ulcerative (Gastrointestinal disorders) | 3 | 1 | 4
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Faecal calprotectin increased (Investigations) | 0 | 1 | 1
Urine protein/creatinine ratio increased (Investigations) | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/90/NCT04074590/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-06): https://cdn.clinicaltrials.gov/large-docs/90/NCT04074590/SAP_001.pdf